CLINICAL TRIAL: NCT03862950
Title: A Double-Blind, Placebo-Controlled Trial of Metformin in Individuals With Fragile X Syndrome (FXS)
Brief Title: A Trial of Metformin in Individuals With Fragile X Syndrome (Met)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: St. Justine's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FXSMET-2018 Version 16
Record Dates: First submitted 2019-02-26; First posted 2019-03-05 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Fragile X Syndrome; Fragile X Mental Retardation Syndrome; Mental Retardation, X-Linked; Genetic Diseases, X-Linked; Trinucleotide Repeat Expansion; Fra(X) Syndrome; Intellectual Disability; FXS; Neurobehavioral Manifestations; Sex Chromosome Disorders
Keywords: Congenital Abnormalities; Metformin; Nervous System Diseases; Chromosome Disorders
MeSH Terms: conditions — Fragile X Syndrome; X-Linked Intellectual Disability; Genetic Diseases, X-Linked; Intellectual Disability; Neurobehavioral Manifestations; Sex Chromosome Disorders; Congenital Abnormalities; Nervous System Diseases; Chromosome Disorders | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo Medication (Placebo Comparator): The placebo will be dosed in a weight-dependent manner. For participants under 50kg at baseline, the initial dose will be 250mg once per day, and if this dose is well tolerated, they will increase each week by 250mg until a maximum dose of 1000mg daily is reached. For participants at and above 50kg at baseline, the initial dose will be 500mg once per day, and if this dose is well tolerated, they will increase each week by 500mg until a maximum dose of 2000mg daily is reached. After the 4-week titration period, each participant will continue dosing at his or her maximum tolerated dose daily for the remaining 12 weeks of the study.
  Interventions: Drug: Placebo Medication
- Active Metformin Medication (Active Comparator): The active metformin medication will be dosed in a weight-dependent manner. For participants under 50kg at baseline, the initial dose will be 250mg once per day, and if this dose is well tolerated, they will increase each week by 250mg until a maximum dose of 1000mg daily is reached. For participants at and above 50kg at baseline, the initial dose will be 500mg once per day, and if this dose is well tolerated, they will increase each week by 500mg until a maximum dose of 2000mg daily is reached. After the 4-week titration period, each participant will continue dosing at his or her maximum tolerated dose daily for the remaining 12 weeks of the study.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Placebo Medication — Placebo liquid or capsules given in parallel to active medication.
  Other Names: Placebo
  Arms: Placebo Medication
Drug: Metformin — Active medication
  Other Names: Glumetza; Glucophage; Fortamet
  Arms: Active Metformin Medication

SUMMARY:
This study is a controlled trial of metformin in individuals with fragile X syndrome between the ages of 6 and 35 years. Participants will be randomized in a double-blind design to either drug or placebo and will attend three visits to the study site in a 4-month period for a series of tests. The primary objectives are to assess safety, tolerability, and efficacy of metformin in the treatment of language deficits, behavior problems, and obesity/excessive appetite in individuals with fragile X syndrome.

DETAILED DESCRIPTION:
This is a multi-center study at the University of Alberta and CHU Sainte-Justine for fragile X syndrome (FXS) patients aged 6 to 35 years inclusive. It is a randomized, double-blind, placebo-controlled trial of metformin (also known as Glumetza, Glucophage, Fortamet), a type 2 diabetes medication that can also improve obesity and excessive appetite.

Metformin has emerged as a candidate drug for the targeted treatment of FXS based on animal studies showing rescue of multiple phenotypes in the FXS model. Metformin may contribute to normalizing signaling pathways in FXS in the central nervous system, which may include activities of mTOR and PI3K, both of which have shown to be pathogenically overactive in FXS. In addition, metformin inhibits phosphodiesterase, which would lead to correction of cAMP levels, and MMP9 production, which is also elevated in FXS. Looking at the potential signaling pathways, metformin appears to be a good candidate for targeting several of the intracellular functions in neurons disrupted in FXS and, therefore, has potential to rescue several types of symptoms in individuals with FXS. Researchers have utilized metformin in the clinical treatment of over 20 individuals with FXS between the ages of 4 and 58 years and have found the medication to be well tolerated and to provide benefits not only in lowering weight gain and normalizing appetite but also in language and behavior. In this controlled trial, the researchers hope to further assess metformin's safety and benefits in the areas of language and cognition, eating and weight loss, and overall behavior.

Each participant will be involved in this trial for a period of 4 months. This will include 3 visits to one of the sites and 5 phone calls. At each visit, the researchers will assess behavioral, cognitive, and language development. The researchers will also assess the side effects of the study medication throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* Subject has Fragile X syndrome with a molecular genetic confirmation of the full FMR1 mutation (>200 CGG repeats) or the other loss of function mutations of the FMR1 gene (SNVs and deletions of the gene).
* Subject is a male or non-pregnant, non-lactating female age 6 through 35 years, inclusive.
* Subjects who are capable of becoming pregnant must use an acceptable method of birth control for the duration of the study. Acceptable forms of birth control include abstinence (only for subjects who are not sexually active), intrauterine devices in place for at least 3 months, oral contraceptives, surgical sterilization, or adequate barrier methods.
* Subject must have a caregiver (parent, guardian, or other legally authorized representative) who is willing to participate in the whole study.
* Subject and caregiver are able to attend the clinic regularly and reliably.
* Subject and/or subject's caregiver is able to understand, read, write and speak English or French fluently to complete study-related materials.
* For subjects who are not their own legal guardian, subject's caregiver is able to understand and sign an informed consent to participate in the study.
* The use of concomitant medication must be stable, in terms of dose and dosing regimen, for at least 4 weeks prior to Screening and must remain stable during the period between first visit (Screening) and the commencement of the study; every effort should be made to maintain stable regimens of allowed concomitant medications from the time of commencement of double-blind study medication until the last study assessment.
* Behavioral/educational treatments must be stable for 4 weeks prior to first visit (Screening) and must remain stable during the period between Screening and the commencement of randomized double-blind study medication.
* 10. Overall age equivalent is not higher than 13 and IQ is not higher than 85, as assessed at Screening on the Leiter-III, and subject must speak at least occasional 3-word phrases.

Exclusion Criteria:

* Families that are not cooperative and will not follow through with the demands of this study.
* Subject has a life-threatening medical problem or other major systemic illness that compromises health or safety and/or would interfere with this study.
* Age younger than 6 or older than 35 years.
* History of intolerable adverse events with metformin.
* Current or recent metformin treatment (within the past 4-months).
* BMI inferior to 2 standard deviations below the mean for age using the World Health Organization scale.
* Serum creatinine > 1.4 mg/dl (female) or > 1.5 mg/dl (male).
* History of metabolic acidosis or a condition with lactic acidosis.
* Severe Vitamin B12 deficiency.
* Pregnancy at screening or unwillingness to use acceptable method of birth control, if applicable.
* Age equivalent higher than 13 or IQ higher than 85 on the Leiter-III at Screening.

Ages: 6 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 125 (Actual)
Dates: Start 2019-05-24 (Actual); Primary Completion 2025-12-16 (Actual); Study Completion 2025-12-16 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Expressive Language Sampling (ELS) mean Number of Different Words (NDW) score | Baseline, End of Treatment/Week 16
  The ELS is collected from shared interactions around a wordless picture book involving the participant and the examiner. The primary outcome measure will be Number of Different Words (NDW) derived from transcripts of audiorecorded samples of spoken language taken from two sampling contexts (conversation and narration), according to procedures described by Abbeduto and colleagues (Abbeduto et al., 1995; Kover et al., 2012). Samples are collected pre- and post- treatment using different books on each occasion. The mean of NDW in conversation and NDW in narration will be computed, and statistically adjusted through analysis of covariance for differences in talkativeness as outlined in Conners et al., 2018. The mean NDW score ranges from 1 to infinite/unspecified. An increase (positive change) in score from baseline to follow-up indicates improvement. The greater the increase, the greater the improvement.

SECONDARY OUTCOMES:
Change from baseline in the FXS-normed Aberrant Behavior Checklist - Community Edition (ABC-C) | Baseline, Week 8, End of Treatment/Week 16
  The ABC-C is a 58-item caregiver-rated behavior scale used to examine treatment effects on challenging behaviors for individuals with FXS in the following domains: (1) irritability, agitation, crying; (2) lethargy, social withdrawal; (3) stereotypic behavior; (4) hyperactivity, noncompliance; and (5) inappropriate speech. Analysis will be performed utilizing the Sansone et al. (2012) FXS-normed ABC scoring measures.
Improvement of symptoms in FXS using the Clinical Impression - Improvement (CGI-I) scale | Baseline, Week 8, End of Treatment/Week 16
  The CGI is a clinician-rated scale utilizing history from the caregiver and incorporating it into a clinical rating, first for severity, and then for clinical follow-up. The CGI-S will be used at the baseline assessment to judge symptom severity as 1 = Normal, not at all ill; 2 = Borderline ill; 3 = Mildly ill; 4 = Moderately ill; 5 = Markedly ill; 6 = Severely ill; and 7 = Among the most extremely ill. The CGI-I will be used at the Week 8 and End of Treatment/Week 16 visits to judge the change in clinical impression as 1 = Very Much Improved; 2 = Much Improved; 3 = Minimally Improved; 4 = No Change; 5 = Minimally Worse; 6 = Much Worse; and 7 = Very Much Worse.
Change from baseline in the Visual Analog Scale (VAS) | Baseline, Week 8, End of Treatment/Week 16
  The VAS will be used to measure the severity of three specific behavioral symptoms targeted in this study: behavior problems, language abilities, and eating behavior. For each behavior the caregiver is instructed to mark their impression of the behavior at the baseline visit and again at the Week 8 and End of Treatment/Week 16 visits. The calculated distance in cm between the visit marks thereby demonstrates whether each behavior stayed the same, improved, or worsened during the study and by how much. The scale is from 0 cm (defined as "worst behavior") to 10 cm ("behavior not a problem").
Change from baseline in the Vineland Adaptive Behavior Scales-Third Edition (VABS-III) Adaptive Behavior Composite Score | Baseline, End of Treatment/Week 16
  The VABS-III is a caregiver survey interview that measures the personal and social skills of individuals from birth through adulthood. It was designed to assess handicapped and non-handicapped persons in their personal and social functioning and is appropriate for individuals of all ages. The Adaptive Behavior Composite (ABC) score is calculated from the caregiver responses using age-adjusted scoring tables. ABC scores range from 20 to 160 and indicate low (20-70), moderately low (70-85), adequate (85-115), moderately high (115-130), or high (130-160) overall adaptive functioning.
Change from baseline in the Anxiety Depression and Mood Screen (ADAMS) overall score | Baseline, Week 8, End of Treatment/Week 16
  The CSHQ consists of a series of questions relating to the sleep habits of children. It will be completed by caregivers of all participants, regardless of participant age, at the baseline, Week 8, and End of Treatment/Week 16 visits.
Change from baseline in the Swanson, Nolan and Pelham Questionnaire (SNAP-IV) overall score | Baseline, Week 8, End of Treatment/Week 16
  The SNAP-IV, based on DSM-V criteria for ADHD, is a caregiver-rated questionnaire that effectively identifies those with and without ADHD and accurately predicts presentation specifier (inattention, hyperactivity/impulsivity, and combined). Its psychometric properties and clinical utility have been demonstrated in multiple studies since its introduction in 2001, and it has been found to be reliable and well validated with normative data from both parents and teachers. It will be completed by caregivers of all participants at baseline, Week 8, and End of Treatment/Week 16.
Change from baseline in the Pediatric Quality of Life Questionnaire (PedsQL) Parent Proxy overall score | Baseline, Week 8, End of Treatment/Week 16
  The PedsQL Parent Proxy consists of a series of questions relating to a child's quality of life and is administered to the caregiver of the participant. The parent proxy module designed for children 8-12 years of age will be administered to the caregivers of all participants, regardless of participant age, because the questions therein are most appropriate for the overall study population's cognitive age and ability. It will be completed at the baseline, Week 8, and End of Treatment/Week 16 visits. For any participants not in school, questions pertaining to "school" will be replaced with references to "work" or other activities in their life.
Change from baseline in the EuroQol-5D (EQ-5D) overall score | Baseline, Week 8, End of Treatment/Week 16
  This is a standardized instrument developed by the EuroQol Group as a measure of health-related quality of life that can be used in a wide range of health conditions and treatments. The EQ-5D consists of a descriptive system and the EQ VAS. We will use the EQ-5D-Y, EQ-5D-Y parent proxy, EQ-5D-3L, and EQ-5D-3L parent proxy depending on the participants age and ability. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale. This can be used as a quantitative measure of health outcome that reflects the patient's own judgement. The scores on these five dimensions can be presented as a health profile or can be converted to a single summary index number (utility) reflecting preferability compared to other health profiles.
Change from baseline in the Care Related Quality of Life (CarerQoL) overall score | Baseline, Week 8, End of Treatment/Week 16
  The CarerQol was designed to measure and value the impact of providing informal care on carers. It combines a subjective burden measure that provides a comprehensive description of the caregiving situation (CarerQol-7D) with a valuation of informal care in terms of well-being (CarerQol-VAS).
Change from baseline in The Memory Game | Baseline, End of Treatment/Week 16
  This is an online test developed in the Bolduc Laboratory done on a tablet at home. Participants are asked to remember association between sets of pictures. The test has been done in typical development and developmental delay for participants 4 years and up. The test has an online consent form followed by a short demonstration video. The participants are then shown pairs of pictures they must remember. Testing is performed right after the presentation and again 24 hours later. For the 24 hours testing, the participants/caregivers will receive an email reminder and will be invited to login to the Memory Game site to perform the association test this time without being shown the demonstration video. The testing takes about 20 minutes the first day and 7 minutes the second day. It will be completed before treatment starts and after treatment ends.
Change from baseline in the Child Sleep Habits Questionnaire (CSHQ) overall score | Baseline, Week 8, End of Treatment/Week 16
  The CSHQ consists of a series of questions relating to the sleep habits of children. It will be completed by caregivers of all participants, regardless of participant age, at the baseline, Week 8, and End of Treatment/Week 16 visits.
Change from baseline in the NIH Toolbox Picture Sequence Memory Test | Baseline, End of Treatment/Week 16
  This test involves recalling increasingly lengthy series of illustrated objects and activities around different themes (e.g., "playing at the park," "working on the farm") that are presented in a particular order on the screen. Encoding, storage, and retrieval of episodic memories depend on a neural network including the temporal lobe (especially the hippocampus), the prefrontal cortex, and limbic/temporal association areas. Patients with FXS perform approximately two standard deviations below normal on PSM, which demonstrates good feasibility, test-retest reliability in both healthy children and those with ID; and moderate correlation with FSIQ.
Change from baseline in the NIH Toolbox Flanker Inhibitory Control and Attention Test | Baseline, End of Treatment/Week 16
  Flanker is a measure of inhibition and visual attention. On each trial, a central directional target is flanked by similar stimuli on the left and right. The participant chooses the direction of the central stimulus. On congruent trials, the flankers face the same direction as the target. On incongruent trials, they face the opposite direction. Patients with FXS demonstrate profound deficits on Flanker, performing about 7 standard deviations below normal, and significantly worse than IQ-matched controls with Down syndrome. This test demonstrates excellent test-retest reliability and correlates significantly with FSIQ and dialing functioning in children and adolescents with ID.
Change from baseline in the NIH Toolbox Dimensional Change Card Sort Test | Baseline, End of Treatment/Week 16
  This is a measure of cognitive flexibility. Two target pictures are presented that vary along two dimensions (i.e., shape and color). Participants are asked to match a series of bivalent test pictures (e.g., yellow balls and blue trucks) to the target pictures, first according to one dimension (e.g., color) and then, after a number of trials, according to the other dimension (e.g., shape). "Switch" trials are also employed, in which the participant must change the dimension being matched. It demonstrates good test-retest reliability and correlates well with FSIQ in children and adolescents with ID, including FXS .
Change from baseline in the NIH Toolbox List Sorting Working Memory Test | Baseline, End of Treatment/Week 16
  This test requires immediate recall and sequencing of different visually and orally presented stimuli. Pictures of different foods and animals are displayed with accompanying audio recording and written text (e.g., "elephant"), and the participant is asked to state the items in size order from smallest to largest, first within a single dimension (either animals or foods, called 1-List) and then on 2 dimensions (foods, then animals, called 2-List). The raw score is the number of items recalled and sequenced correctly.
Change from baseline in the NIH Toolbox Pattern Comparison Processing Speed Test | Baseline, End of Treatment/Week 16
  This test measures speed of processing by asking participants to discern whether two side-by-side pictures are the same or not the same by touching "yes" or "no" (or a happy or frowning face for lower mental age). Participants' raw score is the number of items correct in a 90-second period. The items are designed to be simple to distinguish.
Change from baseline in the NIH Toolbox Oral Reading Recognition Test | Baseline, End of Treatment/Week 16
  The participant is asked to read and pronounce letters and words as accurately as possible. The test administrator scores them as right or wrong. The items are administered by computer adaptive testing (CAT; continuously adapted depending on performance), and participant responses are scored by the examiner. For the youngest children, the initial items require identification of letters (as opposed to symbols) and identification of a specific letter in an array of 4 symbols. A theta score is calculated for this test.
Change from baseline in the NIH Toolbox Picture Vocabulary Test | Baseline, End of Treatment/Week 16
  This measure of receptive vocabulary is administered in a CAT format. The respondent is presented with an audio recording of a word and four photographs on the screen and is asked to select the picture that most closely matches the meaning of the word. A theta score is calculated for this test.
Change from baseline in the NIH Toolbox Speeded Matching Test | Baseline, End of Treatment/Week 16
  This test measures speed of processing by asking participants to discern whether four side-by-side pictures match the target image at the top of the screen. The items are presented one group at a time on the iPad screen, and the participant is given 119.999 seconds of actual presentation time (excluding transitions between items) to respond to as many items as possible (up to a maximum of 130). The items are designed to be simple so as to most purely measure processing speed. Speeded Matching gives a raw score, which is the number of items the participant correctly responds to (up to 130) in 119.999 seconds.
Change from baseline in Eye Tracking | Baseline, End of Treatment/Week 16
  For individuals with FXS, we have demonstrated that the social gaze measure shows decreased visual fixations on the eye region while viewing human faces (with greater fixation to the nose region), and these individuals show abnormal pupillary dilation, an indication of sympathetic nervous system reactivity, compared with controls. While these measures do not appear to map directly onto caregiver-reported anxiety of the individuals level of anxiety, the results are consistent with high rates of social anxiety and sympathetic reactivity in FXS. Stimuli are presented on a Tobii T120 eye-tracker. The system has several benefits that make it conducive to testing individuals with developmental disorders. Stimuli consist of sixty colored photographs of adult human faces each showing a calm, happy, or fearful expression, and sixty scrambled versions of the face images.
Change from baseline in Event Related Potentials during the Auditory Oddball Paradigm and Pseudoword Paradigm | Baseline, End of Treatment/Week 16
  Recently, researchers were able to obtain EEG recordings and ERP responses during an auditory oddball paradigm from patients with FXS enrolled in a controlled trial of minocycline. The study demonstrated the potential feasibility and sensitivity of ERPs as an indicator of cortical processing changes in a targeted treatment trial. It appears to provide a biomarker and measure for the human equivalent of cortical hyperexcitability. Additionally, we will administer a recently developed task looking at EEG habituation to pseudowords to assess word learning with EEG. Data is acquired using a Brainproducts Quickamp system. Raw data is imported into Brainvision Analyzer software for analysis. The continuous data is segmented according to the event type and filtered. We also analyze the EEG data at resting state for the oddball paradigm according to frequency distribution and the occurrence of spontaneous oscillations, and pseudoword habituation with ERP, energy and time-frequency analyses.
Change from baseline in the Sensory Profile-2 or Sensory Profile Adolescents/Adults | Baseline, Week 8, End of Treatment/Week 16
  The Sensory Profile 2 family of assessments evaluates a child's sensory processing patterns in the context of everyday life. The forms are completed by caregivers, who are in the strongest position to observe the child's response to sensory interactions that occur throughout the day. The Adolescent/Adult Sensory Profile was developed to assess sensory processing abilities in individuals beyond childhood. The Sensory Profile Adolescents/Adult is a self report, however, if the participant is unable to complete it themself, we will ask their caregiver to complete it and we will make note of who completed it. The French versions are the Profil sensoriel 2 and the Profil sensoriel-adolescent/adulte.

CONTACTS AND LOCATIONS:
Overall Officials: Francois Bolduc, MD, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - CHU Sainte-Justine, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dy ABC, Tassone F, Eldeeb M, Salcedo-Arellano MJ, Tartaglia N, Hagerman R. Metformin as targeted treatment in fragile X syndrome. Clin Genet. 2018 Feb;93(2):216-222. doi: 10.1111/cge.13039. Epub 2017 Sep 25. PMID 28436599
- [Background] Monyak RE, Emerson D, Schoenfeld BP, Zheng X, Chambers DB, Rosenfelt C, Langer S, Hinchey P, Choi CH, McDonald TV, Bolduc FV, Sehgal A, McBride SMJ, Jongens TA. Insulin signaling misregulation underlies circadian and cognitive deficits in a Drosophila fragile X model. Mol Psychiatry. 2017 Aug;22(8):1140-1148. doi: 10.1038/mp.2016.51. Epub 2016 Apr 19. PMID 27090306
- [Background] Gantois I, Khoutorsky A, Popic J, Aguilar-Valles A, Freemantle E, Cao R, Sharma V, Pooters T, Nagpal A, Skalecka A, Truong VT, Wiebe S, Groves IA, Jafarnejad SM, Chapat C, McCullagh EA, Gamache K, Nader K, Lacaille JC, Gkogkas CG, Sonenberg N. Metformin ameliorates core deficits in a mouse model of fragile X syndrome. Nat Med. 2017 Jun;23(6):674-677. doi: 10.1038/nm.4335. Epub 2017 May 15. PMID 28504725

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-01): https://cdn.clinicaltrials.gov/large-docs/50/NCT03862950/Prot_SAP_008.pdf